CLINICAL TRIAL: NCT03359070
Title: Clinical Study of Non-inferiority (Phase 2), Comparing Dapaconazole (BL123 - Biolab Sanus Farmacêutica Ltda.) Versus Miconazole Nitrate (União Química) in Patients With a Single Lesion of Tinea Cruris.
Brief Title: Clinical Trial Comparing Dapaconazole Versus Miconazole in Patients With Tinea Cruris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galeno Desenvolvimento de Pesquisas Clínicas (Other Government)
Collaborators: Biolab Sanus Farmaceutica (Industry)
Responsible Party: Principal Investigator, Gilberto De Nucci, Doctor, Galeno Desenvolvimento de Pesquisas Clínicas
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GDN 042/13
Record Dates: First submitted 2017-11-27; First posted 2017-12-02 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Tinea Cruris
Keywords: Tinea cruris; dapaconazole; topical antifungal; dermatophytoses
MeSH Terms: conditions — Tinea Cruris; Tinea | interventions — 1-(2-(2,4-dichlorophenyl)-2-(4-(trifluoromethyl)benzyloxy)ethyl)-1H-imidazole; Miconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 - dapaconazole cream 2% (Experimental): Topical application of dapaconazole cream 2%, twice a day (7 to 8 a.m. and 6 to 7 p.m.) for 14 days.
  Interventions: Drug: Dapaconazole
- Group 2 - miconazole cream 2% (Active Comparator): Topical application of miconazole cream 2%, twice a day (7 to 8 a.m. and 6 to 7 p.m.) for 14 days.
  Interventions: Drug: Miconazole Nitrate

INTERVENTIONS:
Drug: Dapaconazole — Application of 1 gram on the lesion.
  Other Names: Zilt
  Arms: Group 1 - dapaconazole cream 2%
Drug: Miconazole Nitrate — Application of 1 gram on the lesion.
  Other Names: Vodol
  Arms: Group 2 - miconazole cream 2%

SUMMARY:
This trial aims to evaluate the efficacy of dapaconazole tosylate 2% cream in the treatment of Tinea cruris compared to the active control miconazole nitrate 2% cream in patients with a single lesion.

DETAILED DESCRIPTION:
This is a phase 2, non-inferiority, monocentric, double-blind, randomized (allocation of treatment), balanced, controlled (active comparator) trial, with two parallel groups.

Randomization depended on inclusion/exclusion criteria, taking into account the confirmation of diagnosis by the direct mycological test and culture performed during the screening phase.

Participants showed up to the clinic, for treatment, during 14 consecutive days, when one of the investigational products (according to the randomization) was applied by a blind member of the study staff. A non-blind member of the study staff weighed the corresponding investigational product and passed on to the blind member only a spatula with the weighed product, in order to maintain the blinded aspect of the trial.

For exploratory purposes, clinical and mycological evaluations was also performed after 7 and after 14 days of treatment.

Safety analysis was performed considering all the randomized patients to which at least one dose of the investigational products has been applied, regardless of the result of the fungal culture.

Conclusion of non-inferiority was based on the per protocol set. It was deemed as per protocol those participants who did not miss more than 20% of the applications and, also, no more than four consecutive application days.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged from 18 to 65 years old, male, or female with no childbearing potential or who are using an effective contraceptive method and who do not plan to become pregnant during the study period.
* Presence of dermatological lesion of Tinea cruris, with an area not exceeding 8 cm², having, also, the diagnosis confirmed by direct mycological (KOH) test and fungus culture.
* No previous treatment with antimycotic medication for the current dermatologic lesion.
* No evidence of other significant diseases, that, at the investigator's discretion, may affect the participation in the clinical trial, in accordance with the protocol requirements.
* Ability to understand the nature and the objective of the clinical trial, including the risks and possible side effects; intention to cooperate with the investigator and act in accordance with the protocol requirements, as confirmed by the informed consent form signature.

Exclusion Criteria:

* Known hypersensitivity to miconazole or to chemically related compounds (azoles) or to the compounds of the investigational products.
* Existing hepatic and/or renal diseases or other pathologic findings, which might interfere with the safety and tolerability of the active ingredients.
* Screening laboratory tests presenting deviations deemed as clinically significant, which, due to possible risks, prevents the participation in clinical trial.
* Treatment, within 3 months prior to the start of the clinical trial treatment, with any drug known to have a well-established toxic potential to major organs.
* Pregnant or lactating women
* Participation in any clinical trial, or intake of any investigational product, within the last six months prior to the inclusion in the clinical trial.
* History of drug addiction.
* Any prior treatment for the present lesion which, at investigator discretion, may interfere with the objectives of the clinical trial.
* Participants who has any condition that prevents him from participating in the study according to the investigator's judgment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2014-01-29 (Actual); Primary Completion 2014-12-10 (Actual); Study Completion 2015-05-06 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with therapeutic cure. | 14 days of treatment
  Proportion of participants, in each treatment group, who achieved therapeutic cure, defined as both clinical and mycological cure, on the assessment performed after 14 days of treatment.
  Clinical cure was considered when there was no more scaling of the lesions, total absence of erythema, itching and desquamation.
  Mycological cure was defined as negative result for the direct mycological examination (potassium hydroxide [KOH] test) and a negative fungal culture.

SECONDARY OUTCOMES:
Number of days until clinical cure | up to 14 days
  Number of days elapsed between the day of start of treatment and the day when the clinical cure was diagnosed, according to the daily assessment, in each treatment group.
Number of adverse events per participant | up to 30 days
  Number of adverse events, in each treatment group, including clinically relevant alterations of vital signs and laboratory tests.

CONTACTS AND LOCATIONS:
Locations (1):
- Galeno Desenvolvimento de Pesquisas Clinicas Ltda. - ME, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No